CLINICAL TRIAL: NCT03386006
Title: Randomized Trial of an Innovative Smartphone Application for Bariatric Surgery
Brief Title: Noom Coach for Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44DK116370 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2017-12-29 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: bariatric surgery; mobile health (mHealth); psychosocial functioning; obesity; weight loss; behavioral activation
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noom Coach for Bariatric Health (Experimental): Self-monitoring will be conducted through Noom Coach for Bariatric Health, and individuals will receive a specialized set of instructions on how to use the app.
  Interventions: Behavioral: Noom Coach for Bariatric Health
- Usual Care (No Intervention): The control group will be a "usual care" condition in which participants are free to seek any assistance for their bariatric surgery care during the study period.

INTERVENTIONS:
Behavioral: Noom Coach for Bariatric Health — Noom Coach for Bariatric Health offers a sustainable, low-cost, coach-led intervention, and an innovative solution to issues with pre-bariatric surgery weight loss. The intervention will take place over 8 weeks.
  Arms: Noom Coach for Bariatric Health

SUMMARY:
The prevalence of overweight in America is a national public health crisis. As more people consider bariatric surgery for the treatment of severe obesity, it is imperative to identify factors influencing surgical outcomes. Technology, particularly the Noom Coach platform, offers a unique opportunity to improve standard interventions utilized in bariatric surgery programs. This study plans to test the efficacy of the Noom Coach platform on patients' adherence behaviors and psychosocial factors compared to standard care.

DETAILED DESCRIPTION:
Overweight and obesity have reached epidemic proportions in the United States. Few behavioral treatments are effective for overweight, and bariatric surgery is consequently an increasingly important option. Although these procedures produce significantly more weight change than psychosocial treatments, post-operative weight losses vary widely, about 20% of patients clearly experience suboptimal weight loss, and a notable subset of these patients demonstrate substantial weight regain. Further, 20-30% report persistence of disturbed eating, depression or anxiety, or impaired health related quality of life. Adherence, or "the extent to which a person's behavior coincides with medical or health advice," contributes to variable weight and psychosocial outcomes, as well as failure to follow dietary guidelines, each of which negatively impacts weight loss.

The present study, utilizing "Noom Coach for Bariatric Health", offers a unique opportunity to overcome obstacles to providing empirically supported treatments and to improve standard interventions utilized in bariatric surgery programs; however, rigorous research on apps is limited, and high-quality, adequately powered, randomized controlled trials with large samples are required. The project will therefore test a combined smartphone app and health coaching system to improve adherence and behavioral outcomes for patients receiving bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in: the Mount Sinai Bariatric Surgery Program and planning to receive a bariatric procedure.
* Between the ages of 18 and 60 at entry to the study.
* Speak English.

Exclusion Criteria:

* Clinically significant cognitive limitations or history of developmental disability.
* History of neurological disorder or injury.
* Current/lifetime Diagnostic and Statistical Manual of Mental Disorders (DSM-5) serious psychiatric disorder, such as bipolar disorder, schizophrenia, or psychotic disorder.
* Acute suicide risk.
* Current DSM-5 alcohol or substance use disorder.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Change in adherence to dietary recommendations | Baseline and 8 weeks
  Change in adherence to recommendations provided within pre-bariatric surgery program will be assessed using the ASA-24 interview. The interview is a 24-hr recall of all food and drink consumed. This interview will serve as the basis for measuring the adherence to dietary recommendations.
Change in adherence to physical activity recommendations (Activity Tracker) | Ongoing
  Change in adherence to physical activity recommendations will be measured using information collected from each participants activity tracker (FitBit). The activity tracker records number of steps taken each day and any physical activity performed.
Change in adherence to physical activity recommendations (IPAQ) | Baseline and 8 weeks
  Change in adherence to physical activity recommendations will also be measured using self reported physical activity using the International Physical Activity Questionnaire (IPAQ) The IPAQ is a 27- item questionnaire that assesses physical activity over the past week as a part of everyday activity, activity as a part of work, and activity as recreation. Scores include both minutes and days spent doing physical activity with higher scores indicating more time spent doing these activities. The measure can be scored categorically (low, moderate, high) or continuously using a defined scoring protocol.

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline and 8 weeks
  Change in EDE-Q at 8 weeks as compared to baseline. Questionnaire to assess for eating disorder symptomology. A 28 item measure with 4 subscales of restraint, eating concern, shape concern, and weight concern. Scores range from 0-168 with higher scores indicating more severe eating disorder pathology. Average scores on each subscale are used in addition to an average global score.
Depression Anxiety Stress Scales (DASS) | Baseline and 8 weeks
  Change in symptoms of depression, anxiety, and stress at baseline and 8 weeks. A 42-item self-report questionnaire assessing three related negative emotional states: depression, anxiety, and stress. Items are scored on a 0-3 Likert scale with ranges within each emotional state for normal, mild, moderate, severe and extremely severe symptoms. Higher scores indicate more severe symptoms. Ranges in severity are reported as sum scores for each emotion state. Depression includes normal (0-9), mild (10-13), moderate (14-20), severe (21-27), extremely severe (28+). Anxiety includes normal (0-7), mild (8-9), moderate (10-14), severe (15-19) extremely severe (20+) Stress includes normal (0-14), mild (15-18) , moderate (19-25), severe (26-33) extremely severe (34+).
Short Form-36 Health Survey (SF-36) | Baseline and 8 weeks
  The SF-36 is a 10-item self-report of health-related quality of life measure that generates eight scaled scored. Individual items are scored 0-100 with higher scores indicating a more favorable health state. The eight subscales, reported as weighted means as (0-100) for each scale, include physical functioning, bodily pain, role limitations due to physical health, role limitations due to personal and emotional problems, emotional well being, social functioning, energy/fatigue, general health perceptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No